CLINICAL TRIAL: NCT03016884
Title: Safety and Tolerability of Herpes Zoster Vaccine in Patients With Rheumatoid Arthritis Immunized Prior to Biologics and Tofacitinib Therapy Initiation
Brief Title: Safety and Tolerability of Herpes Zoster Vaccine Rheumatologic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 142-016-EMC
Record Dates: First submitted 2017-01-01; First posted 2017-01-11 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; anti TNF alpha; tofacitinib; Rheumatoid Arthritis
MeSH Terms: conditions — Herpes Zoster; Arthritis, Rheumatoid | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RA patients (Experimental): RA patients will be administered Zostavax vaccine once 2 weeks before initiation of bDMARD, and be monitored accordingly
  Interventions: Biological: Zostavax vaccine
- Healthy Controls (Experimental): healthy control patients will be administered Zostavax vaccine and be monitored accordingly
  Interventions: Biological: Zostavax vaccine

INTERVENTIONS:
Biological: Zostavax vaccine — After the screening, the eligible patients who provided the informed consent, will be administered the zoster vaccine.
  Other Names: ZOSTAVAX® (Zoster Vaccine Live)

SUMMARY:
The reactivation of varicella zoster virus (VZV) (herpes zoster (HZ)) is of substantial public health concern. Updated ACR recommendations for RA treatment suggest that RA patients aged ≥ 50 years should be vaccinated before receiving biologic or tofacitinib therapy. The Investigators therefore propose a prospective study to evaluate the safety, tolerability, and immunogenicity of a zoster vaccine (Zostavax) in patients with RA, administered at least 2 weeks prior to initiation of anti-TNF biologic and tofacitinib therapy for RA.

This is a 6-week open-label prospective multi-center study evaluating the safety, tolerability, and immunogenicity of Zostavax vaccine in the RA population prior to initiation of biologic/tofacitinib therapy for RA. VZV-specific immune response to vaccine in RA patients will be compared to healthy control subjects ≥ 50 years immunized with Zostavax.

DETAILED DESCRIPTION:
Safety and Tolerability of Herpes Zoster Vaccine in Patients with Rheumatoid Arthritis Immunized prior to biologics and tofacitinib therapy initiation Background The reactivation of varicella zoster virus (VZV) (herpes zoster (HZ)) is of substantial public health concern. Its predilection for the elderly and immunosuppressed make it an important cause of morbidity, causing pain, depression, and long-term disability in the form of post-herpetic neuralgia. The risk of HZ is increased by 1.5 to 2 times in patients with rheumatoid arthritis (RA) compared with the general population.This increase has been attributed to both the underlying disease process and treatments for RA, in particular, corticosteroids, TNFα blocking agents, rituximab, and tofacitinib.

A live attenuated zoster vaccine, administered as a single subcutaneous injection, reduces HZ risk by 70% and 51% among immunocompetent individuals 50 to 59 years and 60 years and older in 2 randomized blinded trials, respectively.

Updated ACR recommendations for RA treatment suggest that RA patients aged ≥ 50 years should be vaccinated before receiving biologic or tofacitinib therapy. Yet, the real world data proves that only minority of RA patients initiating biologic therapy are vaccinated for herpes zoster.

The safety concern is that these individuals may develop varicella infection from the vaccine virus strain. Recently, zoster vaccine safety, tolerability, and immunogenicity were prospectively tested in patients on chronic low-medium dose of corticosteroid therapy. Zoster vaccine was generally well tolerated and immunogenic in this patient population.

Based on the VZV incubation period, the first 42 days following vaccination was chosen as the primary safety risk window in the Shingles Prevention Study, a randomized blinded trial that preceded the FDA approval of the vaccine.

The investigators therefore propose a prospective study to evaluate the safety, tolerability, and immunogenicity of a zoster vaccine (Zostavax) in patients with RA, administered at least 2 weeks prior to initiation of anti-TNF biologic and tofacitinib therapy for RA. The study will specifically focus on the zoster vaccine related adverse events, including injection site reactions, the development of zoster-like lesions, and the rates of clinical herpes zoster.

Study Objective:

1. To evaluate the rate of adverse reactions, injection site reactions, and development of zoster-like lesions following Zostavax administration.
2. To evaluate the rate of clinical herpes zoster events after initiation of biologic and small molecule therapies for RA following Zostavax administration.
3. To evaluate the immunogenicity of Zostavax in RA patients immunized 2 weeks prior to biologic or tofacitinib therapy.

Study Design:

This is a 6-week open-label prospective multi-center study evaluating the safety, tolerability, and immunogenicity of Zostavax vaccine in the RA population prior to initiation of biologic/tofacitinib therapy for RA. VZV-specific immune response to vaccine in RA patients will be compared to healthy control subjects ≥ 50 years immunized with Zostavax.

Healthy volunteers will be recruited from hospital staff and from relatives of patients who agreed to participate in this studyNine Rheumatology Departments across Israel only will participate in the study. These centers are Tel Aviv Medical Center, Sheba Medical Center, Assaf Harofe Medical Center, Shaare Zedek Medical Center, Rabin Medical Center, Bnei Tsion Medical Center, Rambam MedicaL Center, Hahemek Medical center, Carmel Medical Center.

Vaccine Information:

ZOSTAVAX is a lyophilized preparation of live, attenuated varicella-zoster virus (Oka/Merck strain) to be reconstituted with sterile diluent to give a single dose suspension with a minimum of 19,400 PFU (plaque forming units) when stored at room temperature for up to 30 minutes. It is administered as a single subcutaneous injection into the deltoid region of the upper arm.

Study Visits:

Screening Visit/Vaccination The study Investigator will discuss, with each subject, the nature of the study, its requirements, and its restrictions. Written informed consent must be obtained prior performance of any protocol specific procedures. Upon recruitment, patients will be examined by a treating rheumatologist, in order to verify the diagnosis of RA and review the pertinent to vaccination medical history. Patients will be subsequently assessed for RA disease activity.

Procedures to be performed during the screening period include:

Informed Consent Confirmation of RA diagnosis and Classification of RA: subject must have a score of 6 or greater on the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis Medical History as pertinent to HZ vaccination including history of prior and concomitant medications, history of any prior episodes of herpes zoster, and zoster vaccine history.

Assessment of RA activity:

Blood test (ESR, CRP), varicella-zoster virus (VZV) antibody titers by glycoprotein enzyme-linked immunosorbent assay (gpELISA), (will be carried out centrally at tel Aviv Sourasky medical center Immunology laboratory) and future analysis (excluding any genetic tests).

After the screening, the eligible patients who provided the informed consent, will be administered the zoster vaccine.

2- week phone interview based follow up/ Biologic or tofacitinib treatment initiation (etanercept and tofacitinib will comprise 80% of total therapies) At the 2-week visit, vaccine safety will be assessed. Following a two-week interval from the zoster vaccine administration, biologic or tofacitinib treatment will be initiated as scheduled by a treating rheumatologist.

Importantly, no biologic treatment of any kind would be provided by the study project.

4- week phone interview follow up Vaccine safety and adverse effects assessment. 6- week visit Vaccine safety and adverse effects assessment. Assessment of RA activity. Subject Withdrawal Subjects may withdraw from the study at any time at their own request.

Assessments:

Assessment of RA Disease Activity At each study visit, patients will be subsequently assessed for RA disease activity Patient Assessment of Arthritis Pain Patient Global Assessment of Arthritis. Physician Global Assessment of Arthritis Health Assessment Questionnaire - Disability Index (HAQ-DI) Safety Assessment Any adverse reactions/events following zoster vaccine administration will be registered and assessed.

Injection site adverse reactions:

Local pain/erythema/swelling/pruritus/warmth/hematoma/induration Hypersensitivity Post vaccination non-injection-site zoster-like and varicella-like rashes Post vaccination herpes zoster occurrence Systemic adverse reactions Progression/worsening of underlying disease

Adverse effects will be defined according to the following definitions:

MILD Does not interfere with subject's usual function. MODERATE Interferes to some extent with subject's usual function. SEVERE Interferes significantly with subject's usual function.

Blood tests Samples of 15 cc blood only will be taken at two visits: pre-vaccination and post-vaccination (6 weeks). VZV antibody titers will be measured by commercially available ELISA kits.

All data will be deidentified. Only the principal investigator will have access to the table key linking the data sets with personally identifiable information. The study documents will be kept locked at department of rheumatology. The study will be financed by the research funds of the principal investigator.

ELIGIBILITY:
For RA arm:

Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
2. Patients fulfilling the 2010 American College of Rheumatology/European League Against Rheumatism Classification Criteria for RA scheduled for a biologic or small molecule therapy (80% candidates for etanercept or tofacitinib therapies.)
3. Only subjects who are ≥ 50 years old will be administered the zoster vaccine.
4. Subjects who are willing and able to comply with scheduled visits and other study procedures
5. Patients on biologics may participate after a washout period as indicated below :

   1. Etanercept : 2 weeks
   2. Infliximab, Golimumab, Adalimumab : 35 days
   3. Tocilizumab and Abatacept SC : 2 weeks
   4. Tocilizumab and Abatacept IV : 35 days

Exclusion Criteria:

1. History of anaphylactic/anaphylactoid reaction to gelatin, neomycin, or any other component of the vaccine.
2. Previous vaccination with any VZV-containing vaccine.
3. Any type of malignancy, ongoing chemotherapy or radiation therapy.
4. Patients who underwent solid organ transplantation.
5. Patients with AIDS or clinical manifestations of HIV
6. Patients treated with a TNFa inhibitor at the time of recruitment or patients within a year of rituximab administration.
7. Patients receiving daily corticosteroid therapy with a dose ≥10 mg/day of prednisone (or equivalent) for ≥ 14 days and/or methotrexate at the dose above 0.4 mg per kg per week.
8. Patients with an active herpes zoster infection or previous herpes zoster less than 6 months before recruitment.
9. Vaccination with any live vaccine within 4 weeks prevaccination, any inactivated vaccine within 7 days prevaccination, or either during the study period.
10. Blood products transfusion within 5 months prior to vaccination through the study period.
11. Patients with active tuberculosis.
12. History of Guillain-Barre Syndrome

for healthy arm: Inclusion subjects who are ≥ 50 years old will be administered the zoster vaccine.

Exclusion

1. History of past or present autoimmune diseases
2. History or current use of immunosuppressive drugs
3. History of anaphylactic/anaphylactoid reaction to gelatin, neomycin, or any other component of the vaccine.
4. .Previous vaccination with any VZV-containing vaccine.
5. Any type of malignancy, ongoing chemotherapy or radiation therapy.
6. History of underwent solid organ transplantation.
7. Active herpes zoster infection or previous herpes zoster less than 6 months before recruitment.
8. Vaccination with any live vaccine within 4 weeks prevaccination, any inactivated vaccine within 7 days prevaccination, or either during the study period.
9. Blood products transfusion within 5 months prior to vaccination through the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Injection site adverse reactions | 6 weeks
  collecting number of patients with injection site adverse reactions defined as: Local pain/erythema/swelling/pruritus/warmth/hematoma/induration will be assessed by the investigators at follow up visit, and will be asked by phone call.
Number of patients with Hypersensitivity | 6 weeks
  collecting number of patients with hypersensitivity adverse reactions defined as: Any immediate systemic reactions such as anaphylactic reaction, fever, low blood pressure, drug induced rash or urticaria, nausea and vomiting, diarrhea data will be collected at the visit of injection administration, and by phone call 2 weeks past the vaccination
number of patients with Post vaccination non-injection-site zoster-like and varicella-like rashes | 6 weeks
  collecting number of patients with non-injection-site zoster-like and varicella-like rash will be defined as adverse reaction. will be assessed by investigator by phone follow up and at 6 weeks follow up meeting.
Number of patients with Post vaccination herpes zoster occurrence | 6 weeks
  collecting number of patients with Post vaccination herpes zoster occurrence will be defined as adverse reaction. will be assessed by investigator by phone follow up and at 6 weeks follow up meeting.

SECONDARY OUTCOMES:
Immunogenicity measured by varicella-zoster virus (VZV) antibody titers by glycoprotein enzyme-linked immunosorbent assay (gpELISA) | 6 weeks
  of 15 cc blood only will be taken at two visits: pre-vaccination and post-vaccination (6 weeks). Serum will be separated, aliquoted and stored frozen at -20°C until analysis. The serum samples will be stored and tested in the TASMC Laboratory for Arthritis Research. VZV antibody titers will be measured by commercially available ELISA kits. Any other analyses of the serum samples in the future will only be performed after obtaining permission from the institutional ethics committee, as required by law. No genetic test will be performed. The serum samples will not be taken outside of the Tel Aviv Medical Center, unless specific permission is obtained from the institutional ethics committee in the future. Samples of 15 cc blood only will be taken at two visits: pre-vaccination and post-vaccination (6 weeks). Serum will be separated, aliquoted and stored frozen at -20°C until analysis. The serum samples will be stored and tested in the TASMC Laboratory for Arthritis Research. VZV antibody
Tender and Swollen Joint Count (28 joint count) | 6 weeks
  Twenty-eight (28) joints will be assessed by a physician to determine the number of joints that are considered tender/painful. The response to pressure/motion on each joint will be assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial joints). These joints will be further assessed for swelling using the same scale.
  The 28 joints to be assessed are the shoulders, elbows, wrists, metacarpophalangeal (MCP) joints, proximal interphalangeal (PIP) joints, and knees. Artificial joints will not be assessed.
Patient Assessment of Arthritis Pain | 6 weeks
  Participants will assess the severity of their arthritis pain using a 100 mm visual analog scale (VAS) placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponds to the magnitude of their pain.
Patient Global Assessment of Arthritis | 6 weeks
  Participants will answer the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The subject's response will be recorded using a 100 mm VAS
Physician Global Assessment of Arthritis | 6 weeks
  The physician will assess how the subject's overall arthritis appears at the time of the visit. This is an evaluation based on the subject's disease signs, functional capacity and physical examination, and should be independent of the Patient's Global Assessment of Arthritis. The Investigator's response will be recorded using a 100 mm VAS.
Health Assessment Questionnaire - Disability Index (HAQ-DI) | 6 weeks
  The HAQ-DI assesses the degree of difficulty a subject has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities.13 Each activity category consists of 2-3 items. For each question in the questionnaire, the level of difficulty is scored from 0 to 3 with 0 representing "no difficulty," 1 as "some difficulty," 2 as "much difficulty," and 3 as "unable to do". Any activity that requires assistance from another individual or requires the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. The form should then be checked by the site staff for completeness.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Ha'Emek Medical center, Unit of Rheumatology, Afula
  - Carmel Medical Center, Haifa
  - Tel Aviv Medical Center, Unit pf Rheumatology, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smitten AL, Choi HK, Hochberg MC, Suissa S, Simon TA, Testa MA, Chan KA. The risk of herpes zoster in patients with rheumatoid arthritis in the United States and the United Kingdom. Arthritis Rheum. 2007 Dec 15;57(8):1431-8. doi: 10.1002/art.23112. PMID 18050184
- [Background] Schmajuk G, Trivedi AN, Solomon DH, Yelin E, Trupin L, Chakravarty EF, Yazdany J. Receipt of disease-modifying antirheumatic drugs among patients with rheumatoid arthritis in Medicare managed care plans. JAMA. 2011 Feb 2;305(5):480-6. doi: 10.1001/jama.2011.67. PMID 21285425
- [Background] Widdifield J, Bernatsky S, Paterson JM, Gunraj N, Thorne JC, Pope J, Cividino A, Bombardier C. Serious infections in a population-based cohort of 86,039 seniors with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Mar;65(3):353-61. doi: 10.1002/acr.21812. PMID 22833532
- [Background] Yun H, Yang S, Chen L, Xie F, Winthrop K, Baddley JW, Saag KG, Singh J, Curtis JR. Risk of Herpes Zoster in Autoimmune and Inflammatory Diseases: Implications for Vaccination. Arthritis Rheumatol. 2016 Sep;68(9):2328-37. doi: 10.1002/art.39670. PMID 26990731
- [Background] Strangfeld A, Listing J, Herzer P, Liebhaber A, Rockwitz K, Richter C, Zink A. Risk of herpes zoster in patients with rheumatoid arthritis treated with anti-TNF-alpha agents. JAMA. 2009 Feb 18;301(7):737-44. doi: 10.1001/jama.2009.146. PMID 19224750
- [Background] Curtis JR, Xie F, Yun H, Bernatsky S, Winthrop KL. Real-world comparative risks of herpes virus infections in tofacitinib and biologic-treated patients with rheumatoid arthritis. Ann Rheum Dis. 2016 Oct;75(10):1843-7. doi: 10.1136/annrheumdis-2016-209131. Epub 2016 Apr 25. PMID 27113415
- [Background] Schmader KE, Levin MJ, Gnann JW Jr, McNeil SA, Vesikari T, Betts RF, Keay S, Stek JE, Bundick ND, Su SC, Zhao Y, Li X, Chan IS, Annunziato PW, Parrino J. Efficacy, safety, and tolerability of herpes zoster vaccine in persons aged 50-59 years. Clin Infect Dis. 2012 Apr;54(7):922-8. doi: 10.1093/cid/cir970. Epub 2012 Jan 30. PMID 22291101
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Calabrese LH, Calabrese C, Kirchner E. The 2015 American College of Rheumatology Guideline for the Treatment of Rheumatoid Arthritis Should Include New Standards for Hepatitis B Screening: Comment on the Article by Singh et al. Arthritis Care Res (Hoboken). 2016 May;68(5):723-4. doi: 10.1002/acr.22865. No abstract available. PMID 26866816
- [Background] Yun H, Xie F, Delzell E, Chen L, Levitan EB, Lewis JD, Saag KG, Beukelman T, Winthrop K, Baddley JW, Curtis JR. Risks of herpes zoster in patients with rheumatoid arthritis according to biologic disease-modifying therapy. Arthritis Care Res (Hoboken). 2015 May;67(5):731-6. doi: 10.1002/acr.22470. PMID 25201241
- [Background] Koshima I, Higaki H, Soeda S. Combined vascularized fibula and peroneal composite-flap transfer for severe heat-press injury of the forearm. Plast Reconstr Surg. 1991 Aug;88(2):338-41. doi: 10.1097/00006534-199108000-00030. PMID 1852831
- [Background] Singh JA, Furst DE, Bharat A, Curtis JR, Kavanaugh AF, Kremer JM, Moreland LW, O'Dell J, Winthrop KL, Beukelman T, Bridges SL Jr, Chatham WW, Paulus HE, Suarez-Almazor M, Bombardier C, Dougados M, Khanna D, King CM, Leong AL, Matteson EL, Schousboe JT, Moynihan E, Kolba KS, Jain A, Volkmann ER, Agrawal H, Bae S, Mudano AS, Patkar NM, Saag KG. 2012 update of the 2008 American College of Rheumatology recommendations for the use of disease-modifying antirheumatic drugs and biologic agents in the treatment of rheumatoid arthritis. Arthritis Care Res (Hoboken). 2012 May;64(5):625-39. doi: 10.1002/acr.21641. No abstract available. PMID 22473917
- [Background] Russell AF, Parrino J, Fisher CL Jr, Spieler W, Stek JE, Coll KE, Su SC, Xu J, Li X, Schlienger K, Silber JL. Safety, tolerability, and immunogenicity of zoster vaccine in subjects on chronic/maintenance corticosteroids. Vaccine. 2015 Jun 17;33(27):3129-34. doi: 10.1016/j.vaccine.2015.04.090. Epub 2015 May 8. PMID 25964168